CLINICAL TRIAL: NCT06652672
Title: Sentinel Node and Organ-sparing Surgery in Stage I Colon Carcinoma (SENTRY Trial)
Brief Title: Sentinel Node and Organ-sparing Surgery in Stage I Colon Carcinoma
Acronym: SENTRY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meander Medical Center (Other)
Responsible Party: Principal Investigator, Esther Consten, Prof. dr. Esther Consten, Meander Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL84875.100.23; NL84875.100.23 (Other: Medical Research Ethics Committee)
Record Dates: First submitted 2024-10-08; First posted 2024-10-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Colon Cancer; Colon Adenocarcinoma; Sentinel Lymph Node; Sentinel Lymph Node Biopsy; Colon Neoplasms; Colon Neoplasm; Fluorescence; Fluorescence Guided Surgery; Fluorescence Laparoscopy; Fluorescence-guided Resection; Colon Surgery; Indocyanine Green (ICG)
Keywords: Colon cancer; Fluorescence; Sentinel lymph node; Indocyanine green (ICG); Organ sparing surgery; Organ preserving surgery; Local resection
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Multi-center, prospective, non-inferior, partially randomized patient-preference trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Organ-sparing surgery (Experimental): Local resection with sentinel lymph node biopsy
  Interventions: Procedure: Organ-sparing surgery
- Standard of care segmental resection (Active Comparator)
  Interventions: Procedure: Standard of care segmental resection

INTERVENTIONS:
Procedure: Organ-sparing surgery — Endoscopy-assisted laparoscopic/robotic wedge resection and sentinel lymph node biopsy using submucosal injection of ICG.
  Arms: Organ-sparing surgery
Procedure: Standard of care segmental resection — Standard of care segmental resection of the affected part of the colon including removal of regional lymph nodes.
  Arms: Standard of care segmental resection

SUMMARY:
The aim of this study is to reduce the need for colectomy and its' associated morbidity and mortality in patients with pT1-2 colon carcinoma after endoscopic resection and an estimated lymph node metastasis (LNM) risk of >15%, or with macroscopically suspected T1 tumors, by performing an endoscopic-assisted laparoscopic/robotic wedge resection of the tumor or scar, along with sentinel node (SLN) biopsy using indocyanine green (ICG). This intervention will be compared to the standard-of-care segmental resection using a partially randomized patient preference design. The primary outcome is the 3-year recurrence rate.

DETAILED DESCRIPTION:
Colorectal cancer is the third most common type of cancer in the Netherlands and the second leading cause of cancer-related deaths. An increased incidence of T1-2 tumors has been observed following the introduction of population screening programs, leading to more frequent endoscopic excisions. The risk of LNM in T1-2 colon cancers is relatively low. However, local excision does not allow assessment of lymph node status. Moreover, the diagnostic accuracy of computed tomography (CT) and other preoperative imaging modalities for detecting LNM remains limited.

Segmental colonic resections are associated with substantial morbidity. Based on large population-based datasets, 33% of patients experience at least one complication, including anastomotic leakage, with a postoperative mortality rate of 1.5-3.1%. Morbidity is known to substantially impact quality of life and contribute to a high economic burden. Additionally, major symptoms of low anterior resection syndrome (LARS) are present in 21% of patients after segmental resection, with reported effects on quality of life comparable to those experienced by patients who undergo rectal cancer resection and develop LARS.

To minimize unnecessary completion surgery, histopathological risk stratification is applied. In the Netherlands, histopathological risk factors for the presence of LNM in pT1-2 colon cancer are poor (high-grade) differentiation, lymphovascular invasion, high-grade tumor budding (Bd 2-3), and Haggitt level 4. The risk of LNM varies depending on the number of risk factors, pT stage, polyp morphology, and margin status. Completion segmental resection is omitted for pT1-2 tumors with a predicted LNM risk below 15%. Management is guided by risk stratification: for a 5-15% risk, active follow-up is preferred; for a 15-25% risk, active follow-up may be considered as an alternative to completion segmental resection through shared decision-making; and for a >25% risk, segmental resection is the preferred treatment. However, the vast majority of patients with a >15% risk of LNM who undergo surgery experience potential harm but no benefit, as they ultimately do not have LNM. Additionally, suspected T1 tumors are sometimes difficult or impossible to resect endoscopically. In such cases, wedge resection or segmental resection is the standard of care. Depending on T stage and other histopathological risk factors identified after wedge resection, a subsequent segmental resection may still be required. By adding SLN biopsy to the procedure, we aim to avoid the need for segmental resection after wedge resection.

The investigators hypothesize that, in patients who have undergone R0/R1/Rx endoscopic resection of T1-2 colon cancer and have a >15% risk of LNM, or in those with macroscopically suspected T1 tumors, an SLN biopsy combined with wedge resection of the residual tumor or scar can safely spare the majority of patients with negative SLNs from undergoing segmental resection. In our systematic review and meta-analysis, we found a pooled accuracy of 98% and a sensitivity of 80% for SLN detection in T1-2 colon cancer. The investigators use endoscopic submucosal injection of ICG at the tumor site, which carries a low risk of intra-abdominal spillage that could hinder SLN identification.

The SLN biopsy will be combined with an endoscopy-assisted wedge resection of the tumor or scar following endoscopic resection. During the endoscopy-assisted wedge resection, the surgeon first identifies and mobilizes the colon to facilitate the wedge resection. A gastroenterologist then performs a colonoscopy to visualize the scar from the previously resected tumor. With intraluminal endoscopic visualization, the surgeon places a suture to provide traction and position the linear stapler. The gastroenterologist confirms complete inclusion of the scar and ensures lumen patency before the stapler is fired. Endoscopy-assisted limited wedge resection is associated with low complication rates and is performed at lower cost compared to laparoscopic segmental resection. Because no anastomosis is created, the risk of anastomotic leakage is eliminated. This approach could reduce morbidity, mortality, hospital stay, and stoma rates. Although staple line failure and leakage are theoretical risks, such complications have not been reported in previous cases.

Patients with a positive SLN (macro- or micrometastasis) or T3-4 tumors are offered segmental resection. Node-positive patients are recommended to undergo adjuvant chemotherapy if performance status allows. SLN-negative patients do not undergo further surgery and are managed with an intensive follow-up strategy. Assuming 80% sensitivity and a 20% prevalence of lymph node metastasis, the risk of retained positive nodes after SLN biopsy is approximately 4%. Additionally, tumor deposits (TDs) could potentially be missed when patients are treated with SLN biopsy and wedge resection. However, only 0.45% of patients with stage I disease are TD-positive. The investigators consider the absolute risks of missed lymph node metastases and TDs acceptable, given the reduced perioperative morbidity and mortality associated with segmental resection.

The SENTRY trial will be the first to offer organ-sparing surgery combined with an SLN biopsy for patients with selected early-stage colon cancer. This organ-sparing approach is anticipated to improve postoperative mortality, morbidity, hospital stay, quality of life, and costs compared to standard segmental resection, without compromising oncologic outcomes. This multicenter, partially randomized, patient-preference trial will compare the organ-sparing approach with standard-of-care segmental resection to assess oncologic safety.

ELIGIBILITY:
Inclusion Criteria:

* Oral and written informed consent (IC)
* Aged 18 years and older
* Fit for both organ-sparing surgery and colectomy
* Pathologically confirmed T1-2 adenocarcinoma of the colon following R0, R1, or Rx endoscopic resection with an estimated LNM risk >15% (Table 5.2.2. in module 5.2 of the Dutch CRC guideline); or a lesion macroscopically suspected to be (deep-invasive) T1 colon cancer, measuring <40 mm, for which wedge resection is considered the most suitable local resection technique as recommended by the MDT
* The resection scar after local excision is expected to be clearly recognized at endoscopy, either by a tattoo or by detecting a scar in the colorectal segment where no other polypectomies were performed
* Lesion located >25cm from the anus based on endoscopic measurement, or above sigmoid take-off

Exclusion Criteria:

* Patients who opt for active follow-up instead of surgery following shared decision-making
* Distant metastasis
* Lynch syndrome
* Another active malignancy requiring palliative treatment at the time of colon cancer diagnosis
* Previous colorectal cancer within the last 5 years
* Tumours that comprised >50% of the colon circumference before resection
* Tumours involving the ileocaecal valve
* Pregnancy, lactation or a planned pregnancy during the course of the study
* Known allergy to any of the compounds used for SLN identification (ICG, Iodine or Sodium iodide)
* Previous colonic surgery (excluding appendectomy)
* Contra-indication for laparoscopic or robotic surgery
* Severe kidney- or liver failure
* Hyperthyroidism or an autonomously functioning thyroid adenoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2030-12-12 (Estimated); Study Completion 2032-12-12 (Estimated)

PRIMARY OUTCOMES:
3-year recurrence rate | 3 years postoperatively
Successful sentinel lymph node biopsy | Intraoperative
  Percentage of patients undergoing a successful sentinel lymph node biopsy with one or more sentinel lymph nodes detected

SECONDARY OUTCOMES:
5-year recurrence rate | 5 years postoperatively
3-year overall survival | 3 years postoperatively
5-year overall survival | 5 years after postoperatively
90-days complication rate | 90 days postoperatively
  Clavien-Dindo classification
90-days postoperative mortality | 90 days postoperatively
Proportion of patients with preference for standard and experimental treatment, and without preference | 1 day postoperatively
Procedure time of organ-sparing surgery and segmental resection | Directly after surgery, on the same day
Successful wedge resections | Intraoperative
  Percentage of patients undergoing a successful wedge resection
Intraoperative complications | Intraoperative
Upstaging of sentinel lymph nodes due to ultrastaging | During postoperative pathological examination, conducted within two weeks after surgery.
  If sentinel lymph nodes test negative after routine HE staining, ultrastaging is performed. During this process, the lymph nodes are sectioned at 200 µm intervals and examined at three levels using HE staining, as well as immunohistochemistry for cytokeratin AE1/AE3. Sentinel lymph nodes are considered upstaged if they are initially negative on HE staining but are positive during ultrastaging, either with macrometastases (>2 mm) or micrometastases (0.2-2 mm).
Quality of life - EQ5D-5L | From enrollment to the end of study. Questionnaires will be sent preoperatively and 6, 12, 18, 24, 36, 48, and 60 months postoperatively
  EuroQoL 5-Dimension 5-Level. Range 1-5 per dimension. Higher means worse quality of life.
Quality of life - QLQ-CR29 | From enrollment to the end of study. Questionnaires will be sent preoperatively and 6, 12, 18, 24 months postoperatively.
  QLQ-CR29 questionnaire: Organisation for Research and Treatment of Cancer (EORTC) colorectal quality of life module QLQ-CR29. Range 0-100. Higher scores indicate higher levels of symptoms or less functioning.
Quality of life - QLQ-C30 | From enrollment to the end of study. Questionnaires will be sent preoperatively and 6, 12, 18, 24 months postoperatively.
  European Organization for Research and Treatment (EORTC) quality of life questionnaire (QLQ-C30): Range 0-100. A high score on each scale represents a high level in the examined topic, a high score on the global health status for instance represents a high quality of life and a high score in a symptom scale represents a high level of symptoms/problems.
Quality of life - Surv100 | From enrollment to the end of study. Questionnaires will be sent 36, 48, and 60 months postoperatively
  Surv100 questionnaire: European Organization for Research and Treatment (EORTC) quality of life questionnaire survivorship (Surv100). 100 items on a 4- or 7-point Likert scale. A high score on each scale represents a high level in the examined topic, a high score on the global health status for instance represents a high quality of life and a high score in a symptom scale represents a high level of symptoms/problems.
Quality of life - LARS | From enrollment to the end of study. Questionnaires will be sent preoperatively and 6, 12, 18, 24, 36, 48, and 60 months postoperatively
  LARS questionnaire: Low Anterior Resection Syndrome (LARS) score. 0-20 points, no LARS; 21-29 points, minor LARS; 30-42 points, major LARS.
Quality of life - WAI | From enrollment to the end of study. Questionnaires will be sent preoperatively and 6, 12, 18, 24, 36, 48, and 60 months postoperatively
  WAI questionnaire: Work Ability Index. Range 7-49. The total WAI scores are categorized into 4 levels: poor (7-27), moderate (28-36), good (37-43), and excellent (44-49).
Quality of life - iMCQ | From enrollment to the end of study. Questionnaires will be sent 6, 12, 18, and 24 months postoperatively
  iMTA Medical Consumption Questionnaire (iMCQ): The iMCQ includes questions related to frequently occurring contacts with health care providers.
Costs associated with wedge resection and sentinel lymph node biopsy. | 5 years postoperatively
  Bottom-up micro costing will be applied.
Costs standard of care segmental resection | 5 years postoperatively
  Bottom-up micro costing will be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Frank J Voskens, Principal Investigator — Meander Medical Center
Locations (1):
- Meander Medisch Centrum, Amersfoort, Netherlands

IPD SHARING:
Plan to Share IPD: No